CLINICAL TRIAL: NCT03868943
Title: Open Label Safety Study of Solriamfetol to Promote Wakefulness and Improve Cognition and Quality of Life in Patients With Primary Gliomas
Brief Title: Solriamfetol in Improving Sleep in Patients With Grade II-IV Glioma
Acronym: JAZZ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Axsome has conducted a review of the ongoing IST program and are unable to continue supporting this study
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00056700; NCI-2019-01299 (Registry Identifier: National Cancer Institute); P30CA012197 (NIH); CCCWFU 98418 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Solriamfetol (Experimental): Given orally daily
  Interventions: Drug: Soliramfetol

INTERVENTIONS:
Drug: Soliramfetol — Solriamfetol will be dosed by flexible dose titration starting at 75 mg daily in all patients and escalating after 7 days (1 week) to 150 mg daily and then after 7 days to 300 mg daily for a total duration of 3 weeks (flexible dose titration period).

SUMMARY:
This phase II trial studies the side effects of solriamfetol in improving sleep in patients with grade II-IV glioma. Solriamfetol is a wakefulness-promoting drug. Giving solriamfetol may improve sleep, memory, fatigue, mood, or quality of life in patients with brain tumors (gliomas).

DETAILED DESCRIPTION:
Primary Objective:

I. To estimate the safety of solriamfetol at 75 mg daily, 150 mg daily, 300 mg daily as assessed by NCI CTC Adverse Events (v5.0) in patients with primary gliomas compared to prior studies.

Secondary Objective(s):

I. To estimate the effect of solriamfetol on sleep by Epworth Sleepiness Scores (ESS) scores in patients with primary gliomas and compare the effect to previously published scores in patients with OSA

II. To estimate the effect of solriamfetol on sleep quality by Pittsburgh Sleep Quality Index scores

III. To estimate the effect of solriamfetol on neurocognitive function based on a disease-specific neurocognitive battery (see neurocognitive battery below)

IV. To estimate the effect of solriamfetol on patient-reported fatigue (Brief Fatigue Inventory, Cancer Fatigue Scale) & mood (Beck's Depression Inventory)

V. To estimate the effect of solriamfetol on patient-reported QOL (FACT-Br)

VI. To estimate the effect of solriamfetol on objective sleep-wake times by actigraphy and sleep diary (pre- vs post-treatment)

Exploratory Objective(s)

I. To explore a biologic gradient effect of increasing doses of solriamfetol on actigraphy

II. To explore differences in clinical activity of solriamfetol by corticosteroid use, antiepileptic use, and tumor grade.

OUTLINE: This is a dose-escalation study.

Patients receive solriamfetol orally (PO) once daily (QD) for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

WHO Grade 2-4 infiltrating glioma by histologic confirmation

* Where appropriate results from clinically available testing of isocitrate dehydrogenase (IDH) gene mutation status (for all gliomas), chromosome 1p and 19q deletion status (for suspected oligodendrogliomas), and MGMT gene promoter methylation status (for malignant gliomas) must be available in the patient's chart.
* These studies are standard of care molecular studies that are performed as a part of routine clinical practice and allow for integrated molecular subtyping of primary glial tumors.

Epworth Sleepiness Scale (ESS) score >10 within 21 days of enrollment

Clinical and/or radiographic evidence of stable disease within 21 days of enrollment

* Patients must have completed concurrent chemoradiation with recovery of all pre-existing toxicity to CTCAE Grade >1
* Patient who are anticipated to undergo surgery and/or radiation therapy for management of their tumor during the duration of study treatment are NOT eligible.
* Patients who are anticipated to undergo adjuvant chemotherapy are eligible as long as there is no evidence of tumor progression by clinical exam and/or imaging within 21 days of enrollment (see 4.1.2). This determination should be made by clinical documentation and if there is question discussed with the Study Chair. Adjuvant chemotherapy is not an exclusion.
* Patients who are currently undergoing chemotherapy, targeted therapy, immunotherapy, or salvage treatment and have stable disease by imaging are eligible and can continue the current anti-cancer therapy. Patients who will require a new anti-cancer treatment or are anticipated to change anti-cancer treatments are not eligible.

Age > 18 years

Karnofsky performance status ≥ 60%

Life expectancy of greater than 4 months

Patients must have normal organ and marrow function as defined below:

leukocytes >3,000/mcL absolute neutrophil count >1,500/mcL platelets >100,000/mcL total bilirubin 1.5 X institutional upper limits of normal AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal creatinine within normal institutional limits OR creatinine clearance >50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

* The effects of solriamfetol on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Receiving active radiation therapy (including patients who are within 28 days of completing radiation therapy)
* Anticipated to undergo radiation therapy or require neurosurgical intervention during the period of active treatment(i.e. within the next 4 months)
* Contraindication to solriamfetol based on drug-drug interactions or concurrent systemic illness that precludes drug treatment
* Patients who have not recovered to < CTCAE grade 2 toxicities related to prior or current therapy are ineligible.
* Exception for laboratory-based or other adverse event that is stable and not anticipated to interfere with study related treatment must be reviewed and approved by the study chair
* Customary bedtime later than midnight
* Known and/or documented history of obstructive sleep apnea (OSA)
* Uncontrolled behavioral or psychiatric disorder (including suicidal ideation)
* Current excessive caffeine use (> 600 mg/day or > 6 cups of coffee/day)
* Current or prior history of alcohol or drug abuse within the last 2 years as assessed by the treating clinician
* Nicotine dependence that is currently interfering with sleep based on assessment by the treating clinician
* Concurrent use of selective serotonin or norepinephrine reuptake inhibitors (e.g. selective serotonin reuptake inhibitor [SSRI], serotonin and norepinephrine reuptake inhibitors [SNRI]) within 14 days of study enrollment
* Patients who are currently taking these agents may be tapered at the direction of the treating physician prior to study enrollment
* Patients taking other medications such as narcotics, benzodiazepines, antipsychotics, antiepileptics, corticosteroids, or over-the-counter sleep aids can be enrolled. It is recommended that the doses of these medications remain the same throughout the portion of active study treatment unless there is a medical indication for dose adjustment which will be determined by the treating physician
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to solriamfetol
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with solriamfetol, breastfeeding should be discontinued if the mother is treated with solriamfetol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated early. Only 2 participants were enrolled in this study, with only one completing fully. Based on the low enrollment number, some outcomes have no data reported while other outcomes are reported in broad ranges in order to protect and maintain participant privacy/confidentiality.
Period: Overall Study
Arm/Group | Solriamfetol
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Solriamfetol
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  45-70 years | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  White male | 1
  White female | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion With Grade 3 or Higher Adverse Events
Description: National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be used for scoring toxicity and adverse events. Score of 1 to 5 (1 = mild, 5 = death). The proportions of subjects who experienced grade 3 or above toxicities will be estimated
Time Frame: Duration of treatment (timing ranges from 3 weeks to 9 weeks past start of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Epworth Sleepiness Scale
Description: The effect of solriamfetol on patient-reported sleep using Epworth Sleepiness Scale measuring how likely participants are likely to doze off or fall asleep in certain situations (8 situations), in contrast to feeling tired. Scale of 0 would never doze, 1 - slight chance of dozing, 2 - moderate chance of dozing and 3 - high chance of dozing. Score is the sum of the eight items (range 0-24)
Time Frame: End of treatment (timing ranges from 3 weeks to 9 weeks past start of treatment)
Population: The study was terminated early with only 2 participant were enrolled in this study. Based on the low enrollment number, data is reported in broad ranges in order to protect and maintain participant privacy/confidentiality.
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol
Number analyzed (Participants) | 2
Participants
  ESS total score 0-2 | 0
  ESS total score 2-18 | 2
  ESS total score 19-24 | 0

3. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. Each item is on a scale 0 - 3. The total score is a sum of the seven items, ranging from 0-21 with lower scores indicating better sleep.
Time Frame: End of treatment (timing ranges from 3 weeks to 9 weeks past start of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol
Number analyzed (Participants) | 2
Participants
  PSQI total score 0-5 (good sleep quality) | 0
  PSQI total score 6-21 (bad sleep quality) | 2

4. Secondary Outcome: Neurocognitive Battery Record
Description: Evaluation of attention, concentration, information processing speed, learning/memory and aspects of higher-order executive functions to be done at baseline and end of treatment only.
Time Frame: post treatment
Population: The study was terminated early with only 2 participant were enrolled in this study with only one patient completing the neurocognitive battery at the conclusion of the treatment. Since data for only one patient is available, no results are reported to protect the privacy of the patient.
Arm/Group | Solriamfetol
Number analyzed (Participants) | 0

5. Secondary Outcome: Cancer Fatigue Scale (CFS)
Description: 15-item self-administered patient-reported questionnaire exploring both overall and domain specific fatigue in cancer patients. The instrument explores three fatigue domains: physical effects of fatigue, cognitive effects, and affective issues related to cancer fatigue. Each response is measured 1 - No, 2 - a little, 3 - somewhat, 4 considerably and 5 - very much, with a sum of the 15 items as the total score (range 15-75). Higher scores generally indicate greater fatigue/severity.
Time Frame: End of treatment (timing ranges from 3 weeks to 9 weeks past start of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol
Number analyzed (Participants) | 2
Participants
  CFS total score 15-35 | 2
  CFS total score 36-55 | 0
  CFS total score 56-75 | 0

6. Secondary Outcome: Beck's Depression Inventory (BDI)
Description: A 21 item self-scored questionnaire to assess levels of depression. Each item is rated on a scale from 0-3, with the total score being the sum of the 21 items (range 0-63).
Time Frame: End of treatment (timing ranges from 3 weeks to 9 weeks past start of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol
Number analyzed (Participants) | 2
Participants
  BDI score 0-40 (none - severe depression) | 2
  BDI score 41-63 (Extreme depression) | 0

7. Secondary Outcome: FACT-Brain Module (FACT-Br)
Description: An instrument measuring general quality of life (QOL) that reflects symptoms or problems associated with brain malignancies across 5 scales (physical well being, social/family well being, emotional well being, functional well being and additional concerns). Each of the 50 items are on a scale: 0 - not all all, 1 - a little bit, 2 - somewhat - 3 - quite a bit and 4 - very much. Total score has a range 0-200. Higher scores across all subscales and total scores indicate a better quality of life
Time Frame: End of treatment (timing ranges from 3 weeks to 9 weeks past start of treatment)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Solriamfetol
Number analyzed (Participants) | 2
Participants
  0-80 | 0
  81-160 | 2
  161-200 | 0

8. Secondary Outcome: 7 Day Actigraphy
Description: Actigraph devices are worn on the wrist for 7 days and record movements that can be used to estimate sleep patterns using specialized computer software programs. Completion of actigraphy will be done from baseline to end of treatment and recorded with the sleep-diary data.
Time Frame: Approximately over 10 weeks post treatment
Population: The study was terminated early and this data was not collected at the end of study treatment due to patient refusal.
Arm/Group | Solriamfetol
Number analyzed (Participants) | 0

9. Secondary Outcome: 7-day Patient-Reported Sleep Diary
Description: Participants will be provided a sleep diary at the time of consent and/or study enrollment. All sleep diaries will be collected over 7-days including at pre-study baseline, throughout each dose of the dose escalation phase, and during the first 7-days and last 7-days of the fixed dose drug continuation phase of the study. Caregivers may complete sleep diaries for patients.
Time Frame: Approximately 10 weeks post treatment
Population: The study was terminated early and this data was not collected at the end of study treatment due to patient refusal.
Arm/Group | Solriamfetol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 months.
Arm/Group | Solriamfetol
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solriamfetol (N=2)
Other (Gastrointestinal disorders) | 2 (6)
Other (Infections and infestations) | 1 (1)
Other (Nervous system disorders) | 1 (1)
Other (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT03868943/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT03868943/ICF_000.pdf